CLINICAL TRIAL: NCT02212535
Title: Open Study of Phase I / II Evaluating Tolerance and Efficacy of Mobilization and Collection of Peripheral Hematopoietic Stem Cells Device After a Single Injection of 0.24mg/kg of Plerixafor in Sickle Cell Patients
Brief Title: Assessment of Tolerance of Mobilizing Peripheral Hematopoietic Stem Cells by Plerixafor in Sickle Cell Patients
Acronym: DrepaMob
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAO13017; 2014-001650-42 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Major Sickle Cell Syndrome of Type SS or Sβ Thalassemia
Keywords: Sickle cell disease; Open monocenter study; Phase I/II; hematopoietic stem cells; Plerixafor
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor (Experimental): Adult patients affected by major sickle cell syndrome (SS or Sβ thalassemia)
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — 0.24 mg / kg / day, by subcutaneous injection, 11h before the beginning of cytapheresis

SUMMARY:
The purpose of this study is to assess the tolerance and efficacy of mobilizing hematopoietic stem cells after a single injection of plerixafor (0.24mg/kg) in 3 adult patients (or 5, if results of the first 3 patients are not reproducible) affected by sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is a genetic disorder caused by a point mutation in the coding region of the gene of beta-globin with the consequence the production of an abnormal (betas-globin). This mutation is responsible for the polymerization of deoxygenated HbS chains. Polymers make red blood cells (RBC) rigid, and change their shapes and are responsible of structural lesions of the membrane, altering the rheological properties of the RBC and altering blood flow of microcirculation. The two ultimate consequences of all these changes are intravascular haemolysis and the occurrence of vaso-occlusive episodes. Allogeneic hematopoietic stem cells (HSC) transplantation is the only curative treatment for these patients, but only 25% of them have a HLA-genoidentical family donor. In the absence of a compatible donor, gene therapy with model autograft could be a valid alternative. However, gene therapy for the curative treatment of sickle cell disease requires an optimal number of genetically modified HSC to reinject the patient. In contrast to beta-thalassemia patients, the mobilization of HSC in peripheral blood by growth factors such as G-CSF in patients with sickle cell can trigger a vaso-occlusive crisis.

The onset of action of plerixafor is very fast. In pharmacodynamic studies in healthy volunteers, mobilization peak of CD34 + cells was observed between 6 and 9 hours after administration of plerixafor. One injection per day for 1 to 2 days should be sufficient to achieve an optimal collection (unlike the 5-6 days required for mobilization of HSC in G-CSF used as the only growth factor). The duration of exposure to risk is thereby theoretically reduced.

We propose an drug test - Phase I/II trial - monocenter- non-comparative - not randomized - uncontrolled - Open.

In this protocol, we propose to assess the safety and efficacy of peripheral HSC mobilization in three major sickle cell patients (SS or Sbeta thalassemia) (or five, if results of the first 3 patients are not reproducible) by a single injection of plerixafor after significant decrease of HbS rate. Adequate number of CD34 + cells collected will be a key point in the success of possible and subsequent autologous graft of genetically modified HSC; a dose> 3.106 cells / kg CD34 + is necessary. Mobilized and collected cells will be stored for a possible future gene therapy or as not handled backup graft.

These three patients will be included sequentially; new inclusion will take place only if no serious adverse events have occurred in patients being participated in the trial. Recruitment will take place during the consultation in Apheresis Therapeutic Unit / Department of Biotherapy at the Necker-Enfants Malades Hospital. Patients being recruited from the cohort of adults with sickle cell disease at the Hospital Necker-Enfants Malades, the principal investigator will have seen the patient in consultation in the weeks preceding the decision to propose him to take part in research. This consultation will constitute within the framework of this protocol, prior medical examination.

Before plerixafor injection, the patient will be subjected to one or more red cell exchange order to reduce the post-transfusion HbS rate to less than 30% and if possible around 15%. If the patient is under treatment with hydroxyurea, it will be stopped 3 months before collecting peripheral HSC and replaced by an exchange transfusion to the rhythm of once per month.

If the patient is not under treatment with hydroxyurea, he will have only 2 or 3 exchange transfusions during the month before collecting peripheral HSC.

Treatment with plerixafor will be administered in the Adult Intensive Care Unit of the Necker - Enfants malades Hospital. He/She will be under scope, will receive oxygen therapy and hyperhydration (physiological saline per day); his/her ionogram and phosphatemia will be monitored. The procedures of mobilization and collection by apheresis peripheral HSC will be performed by the haematologist doctor and a specialist nurse. The HSC's collection will be made in Apheresis Therapeutic Unit. A member of the LTCG team will retrieve samples in intensive care and will provide their transport to the laboratory for possible transformation. The patient will remain hospitalized after collection of peripheral HSC under the same conditions of treatment and monitoring (scope, oxygen, hyperhydration) until the number of White Blood Cells remain lower than 10x10^9 / L or new income at their count base. HSB's collection and related hospitalisation will be performed according to JACIE (Joint Accreditation Committee of ISCT-EBMT) program and subsequent Standard Operating Procedures in force both at Clinical Unit and Laboratory of Cell and Gene Therapy (LTCG) of the Department of Biotherapy.

The dispensation of treatment will be performed by the Internal Use Pharmacy (PUI) of the Necker-Enfants malades Hospital. Specific prescriptions of plerixafor from the study will be made available to the investigators.

A total of 15 visits for patients with hydroxyurea at screening, and 12 visits for patients without hydroxyurea (including final visit) are scheduled for this trial. The total study duration is 24 months, the duration of inclusion is 14 months.

The data required for the analysis of the study will be reported in a paper case report forms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Affiliated or beneficiary of a health insurance regimen
* For women of childbearing age, not pregnant and use effective contraception during the entire participation in research.
* Affected by a major sickle cell SS or Sβ thalassemia whose diagnosis must have been confirmed by a study of hemoglobin.
* Have the potential indication of allogenic bone marrow and don't have identical-HLA siblings.
* Have a general condition corresponding to a functional index of Lansky ≥ 80%
* Have been treated and followed for at least the previous two years in a specialized center where they got a full assessment of their disease
* In addition to the general eligibility criteria, sickle cell patients must have one or more of the following risk factors despite hydroxyurea treatment with for at least 4 months, except in cases of bad tolerance to hydroxyurea:

  * Severe recurrent vaso-occlusive episodes of duration > 48 hours or having required hospitalization for more than 24 hours (defined by at least two episodes during the previous year or in the year preceding the setting up of regular transfusion protocol)
  * And /or recurrent Acute Chest Syndrome (at least 2 episodes) - defined by the presence of a new pulmonary infiltration involving at least one complete pulmonary segment (but excluding atelectasis) with chest pain and/or fever (> 38 5), and / or tachypnea, and / or wheezing or cough without infectious syndrome
  * Osteonecrosis of 2 or more joints.
  * Anti-erythrocyte alloimmunization (>2 antibodies).
  * Presence of sickle cell cardiomyopathy documented by Doppler echocardiography.
* Informed and signed consent

Exclusion Criteria:

* Patient who to his knowledge and that of the investigator, is unable to follow the visits required by the protocol
* Any form of disorder that, according to the investigator, may compromise the ability of the patient to give an informed written consent and / or to conform to all required procedures of the study.
* Positive serology for HIV-1/2, HTLV-1/2, syphilis, HCV and / or HBsAg
* Bacterial, viral, fungal or parasitic active infection with clinical signs requiring hospitalization for more than 24 hours
* Recurring Malaria
* Personal history of cancer, myeloproliferative hematopathy or immune deficiency
* Cerebral vasculopathy highlighted by transcranial Doppler ultrasound or pathological MRI
* Heart failure and / or heart rhythm disorder and / or myocardial infarction
* History of allogeneic graft of hematopoietic stem cells
* Diagnosis of a psychiatric disorder that could compromise his/her ability to participate in the study
* Current Pregnancy or breastfeeding
* For women of childbearing potential no use effective contraception throughout the whole treatment duration
* Major dysfunction of :

  * Liver : transaminases superior or egal at 3 times more than normal
  * Heart with alteration of the left ventricular ejection fraction (LVEF)
  * Pulmonary High blood pressure confirmed by catheterization
  * Renal with calculated clearance with of creatinine < 30%
  * Severe iron overload with abnormal cardiac T2* MRI < 10 ms
  * Lung with level of oxygen saturation <90% (outside times of crisis) or DLCO < 60% in the absence of infection
* Current participation in another interventional clinical trial
* Polynuclear superior or egal at 10.000/mm3 to the base state without infection or inflammatory syndrome
* Patient under Medical Assistance State
* Patient under guardianship
* Hypersensitivity to plerixafor or any excipient contained in MOZOBIL®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Complication of disease | Day 0 until Month 6 post treatment
  Clinical examination

SECONDARY OUTCOMES:
Efficacy of HSC mobilization | Day 1
  Assessed by the Rate of circulating CD34+
Evaluation of HSC collection | Day 1
  Apheresis

CONTACTS AND LOCATIONS:
Overall Officials: Jean - Antoine RIBEIL, MD, PhD, Study Director — Hôpital Necker - Enfants Malades, Public Hospitals of Paris
Locations (1):
- Hôpital Necker - Enfants Malades, Paris, France

REFERENCES:
- [Background] Lagresle-Peyrou C, Lefrere F, Magrin E, Ribeil JA, Romano O, Weber L, Magnani A, Sadek H, Plantier C, Gabrion A, Ternaux B, Felix T, Couzin C, Stanislas A, Treluyer JM, Lamhaut L, Joseph L, Delville M, Miccio A, Andre-Schmutz I, Cavazzana M. Plerixafor enables safe, rapid, efficient mobilization of hematopoietic stem cells in sickle cell disease patients after exchange transfusion. Haematologica. 2018 May;103(5):778-786. doi: 10.3324/haematol.2017.184788. Epub 2018 Feb 22. PMID 29472357